CLINICAL TRIAL: NCT03082963
Title: Mapping Electrogram Morphology Recurrence for Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Goldberger (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey Goldberger, Chief, Cardiovascular Division, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150757; 1R41HL127907-01A1 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-17 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EMR Feasibility (Other): In this feasibility study, all ten patients will undergo EMR mapping which will be used to guide ablation.
  Interventions: Device: Electrogram Morphology Mapping (EMR)

INTERVENTIONS:
Device: Electrogram Morphology Mapping (EMR) — Fifteen second AF recordings will be made using a multipolar electrode catheter to map the entire right atrium & then the left atrium.

SUMMARY:
The overall goal of this project is to test the feasibility of performing real-time electrogram morphology recurrence (EMR) mapping in patients with persistent atrial fibrillation (AF) to locate areas of high electrogram morphology recurrence rate. The Investigator believe that the EMR mapping can be integrated into cardiac mapping and used to identify potential sites for ablation. Furthermore, this study could help demonstrate the efficacy of this technology's ability to terminate or slow AF.

The Investigator will test this technology on ten subjects undergoing a second ablation procedure. The Investigator will map the AF utilizing the EMR to indicate locations of stable activity and ablate the area. The Investigator believes that the study could produce acute AF termination or AF cycle length slowing. In addition to testing the real-time electrogram morphology recurrence mapping, the study would also like to determine the acute effects of radiofrequency ablation of areas of high recurrence rates and determine long term freedom from AF following ablation of areas of high recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Male and female at least 21 years of age
* persistent Afib with one prior failed ablation for persistent or long standing persistent Afib

Exclusion Criteria:

* Inability to sign consent
* Patients with a life expectancy less than one (1) year
* Patients with chronic kidney disease with sufficiently low GFR that precludes either CT angiogram of the heart or contrast MRI study
* Pregnant women and women that are breast feeding
* Patients with multiple (2 or more) prior failed ablations
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Mitrani, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EMR Feasibility
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EMR Feasibility
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Real-time Electrogram Morphology Recurrence (EMR) Mapping Feasibility
Description: As measured by number of patients where real-time EMR mapping is completed.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | EMR Feasibility
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Ablation Acute Effects
Description: ablation based on EMR map as measured by number of participants that terminate atrial fibrillation.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | EMR Feasibility
Number analyzed (Participants) | 10
Participants | 0

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events will be measured by the type of adverse event, severity, and whether the AE/SAE is related to the mapping
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | EMR Feasibility
Number analyzed (Participants) | 10
Participants | 2

4. Secondary Outcome: Ablation Acute Effects
Description: ablation based on EMR map as measured by number of participants that slow atrial fibrillation cycle length by at least 15%.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | EMR Feasibility
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | EMR Feasibility
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMR Feasibility (N=10)
Post ablation procedure -Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMR Feasibility (N=10)
Pain from blood pressure cuff (Injury, poisoning and procedural complications) | 1 (1) — Pain from blood pressure cuff in the left upper extremity during procedure
Exacerbation of congestive heart failure (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03082963/Prot_SAP_000.pdf